CLINICAL TRIAL: NCT06611657
Title: Anlotinib Hydrochloride Combined With Whole Brain Radiotherapy for the Treatment of Brain Metastases in Small Cell Lung Cancer
Brief Title: Antirotinib Hydrochloride Plus Whole Brain Radiotherapy for Small Cell Lung Cancer With Brain Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2766
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Whole Brain Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib hydrochloride (Experimental): Subjects received antirotinib hydrochloride capsules, 1 capsule (12mg) once a day.
  Interventions: Drug: Antirotinib hydrochloride

INTERVENTIONS:
Drug: Antirotinib hydrochloride — Oral antirotinib treatment was started 2 weeks before radiotherapy for brain metastases, stopped for 1 week after 2 weeks, and continued after radiotherapy until tumor progression
  Other Names: Anlotinib hydrochloride + Brain radiotherapy

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of whole brain radiotherapy combined with antirotinib hydrochloride in the treatment of brain metastases in small cell lung cancer

DETAILED DESCRIPTION:
This was a single-center, single-arm trail. Enrolled patients were pathologically diagnosed with small cell lung cancer and had completed at least 4 cycles of first-line chemotherapy. Patients with brain metastases at first visit or during treatment were treated with whole brain radiotherapy combined with anlotinib hydrochloride. Oral antirotinib was started 2 weeks before radiotherapy for brain metastases and stopped for 1 week after 2 weeks. After radiotherapy, antirotinib was continued until tumor progression. Efficacy and toxicity data were collected for evaluation and analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Small cell lung cancer confirmed by pathology, completion of at least 4 cycles of first-line chemotherapy, and measurable disease according to RECIST criteria.
2. The expected survival time is more than 3 months.
3. Intracranial metastases ≤10.
4. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Patients who have used antiangiogenic drugs within the previous 1 month.
2. Non-small cell lung cancer (including small cell carcinoma and non-small cell carcinoma mixed lung cancer).
3. Small cell lung cancer with hilar invasion or hemoptysis.
4. Patients with intracranial acute, subacute cerebral infarction, intracranial lesions acute, subacute hemorrhage.
5. An unresolved acute toxic reaction period higher than grade 2 of CTC-AE(4.0) due to any prior treatment.
6. Advanced patients with severe symptoms, tumors that have spread to the internal organs, and a short-term risk of life-threatening complications.
7. Patients with life-threatening conditions of other severe and/or uncontrolled diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression-free survival | 6 months
  Time from enrollment to intracranial tumor progression or death

SECONDARY OUTCOMES:
Overall Survival | 1 year
  The time from enrollment to death from any cause was calculated as the time of death. For participants who were lost to follow-up, the time of death was usually the time of the last follow-up.
progression-free survival | 6 months
  The time from enrollment to tumor progression (any aspect) or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Lei Deng, MD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No